CLINICAL TRIAL: NCT05698979
Title: Evaluation of Botulinum TOXin Type a in the Treatment of Buerger's Disease
Acronym: BETOX
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/20/0445
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Buerger Disease; Raynaud Syndrome
Keywords: botulinum toxin A; botox; feasibility; raynaud; buerger; tolerance
MeSH Terms: conditions — Thromboangiitis Obliterans; Raynaud Disease | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- drug administration (Experimental): Botox Injection
  Interventions: Drug: BOTOX INJECTION

INTERVENTIONS:
Drug: BOTOX INJECTION — The patient will be treated with a single session with botulinum toxin A injections at the hospital, and the judgmental criteria will be assessed at 1, 3 and 6 months post injections.
  The injections will be made in 4 injection points at the palmar or distal plantar fold, at the level of the neurovascular beams, 2h after topical anesthesia by lidocaine cream under occlusion, associated or not with nitrous oxide inhaled at the time of the injections (BOTOX® 100 U).
  In the event of multiple lesions, a single limb is injected based on clinical severity (ulcer, gangrene) and ischemia parameters (lowest TCPO2).
  Other Names: botulinum toxin

SUMMARY:
The main objective is to assess the feasibility of treatment by injecting botulinum toxin A into the hand or foot of patients with signs of critical ischemia secondary to Buerger's disease. The injection of botulinum toxin A is carried out at the end of a single session during an hospitalization. Furthermore, tolerance and effects on the disease are evaluated at 1, 3 and 6 months post injections.

DETAILED DESCRIPTION:
Buerger's disease or obliterate thromboangiitis(TAO) is a rare disease. It is an inflammatory, segmental and occlusive disease affecting small and medium caliber arteries and veins in the extremities of the limbs. It mainly affects young men, who traditionally smoke, before the age of 45. There is currently no specific treatment for Buerger's disease. Surgical treatment is rarely feasible, due to distal and diffuse damage. Several studies have evaluated the perivascular injection of botulinum toxin type A (BTX) in patients with severe Raynaud syndromes linked to scleroderma, with promising results.

Studies with BTX have shown reduced pain, improved tissue perfusion with laser doppler, and healing of digital ulcers.

The patients are treated with a single session with botulinum toxin A injections during an hospital visit, and the judgmental criteria are assessed at 1, 3 and 6 months post injections.

The injections are made at 4 injection points at the palmar or distal plantar fold, at the level of the neurovascular beams, 2h after topical anesthesia by lidocaine cream under occlusion, associated or not with nitrous oxide inhaled at the time of the injections (BOTOX® 100 U, botulinum toxin A injections in each hand or foot, for a final dose of 50 U (1 ml) per extremity).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. patient with Buerger's disease according to Olin criteria (ref)
3. with digital ischemia with critical upper or lower limb ischemia criteria defined as Upper limb: pain and/or trophic disorders for at least 15 days AND digital pressure less than 50 mmHg Or TCPO2 30 mmHg) Or/and Lower limb: pain and/or trophic disorders for at least 15 days AND ankle pressure less than 50 mmHg (70 mmHg if diabetes), or 30 mmHg at the toe (50 mmHg if diabetes) or TCPO2 30 mmHg).
4. Ability to attend study visits
5. Ability to complete daily study agenda
6. Ability to give free and informed consent
7. Membership of a Social Security scheme

Exclusion Criteria:

1. History of myasthenia gravis or Eaton-Lambert syndrome
2. History of inflammatory myositis for less than 2 years or pre-existing motor neuron disease or superior limb neuropathy.
3. Known allergy to botulinum toxin or cream lidocaine, albumin or inhaled nitrous oxide/oxygen.
4. Progressive infection of one hand or foot
5. Aminoglycoside treatment
6. Pregnant or nursing women
7. History of vascular surgery of surgical sympathectomy of upper or lower limb
8. Revascularization procedure considered within 3 months of inclusion
9. Risk of major amputation within 3 months of inclusion
10. Iloprost expected within one month of study treatment
11. Hyperbaric chamber sessions scheduled within one month of study treatment
12. Life expectancy less than 6 months
13. Contraindication to one or more of the following products: BOTOX 100 UNITS ALLERGAN, LIDOCAINE/PRILOCAINE 5%, cream or NITROUS OXIDE MEDICINAL
14. Patients treated by class III anti arhythmic drugs for example amiodarone 15 ) Patient with guardians, curators, or protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility in Number of patients | through study completion, an average of 18 months
  The feasibility criterion corresponds to the number of patients who actually received the planned injections within the defined time limits, among the patients who should have received the injection according to the criteria of the protocol.

SECONDARY OUTCOMES:
tolerance of participants | during injection
  collection of temporary low grade adverse events (hematoma, erythema, ecchymosis at the injection site, pain, before/after and during injection)
tolerance of participants | 2 hours after injection
  collection of temporary low grade adverse events (hematoma, erythema, ecchymosis at the injection site, pain, before/after and during injection)
tolerance during injection | during injection
  collection of temporary high grade adverse events (muscle weakness, temporary or prolonged headache, general muscle weakness or muscle group at distance from injection site, difficulty swallowing, dyspnea, immediate allergic reaction to injections)
tolerance after injection | 2 hours after injection
  collection of temporary high grade adverse events (muscle weakness, temporary or prolonged headache, general muscle weakness or muscle group at distance from injection site, difficulty swallowing, dyspnea, immediate allergic reaction to injections)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Malloizel-Delaunay, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/AOMI_recos.pdf